CLINICAL TRIAL: NCT02255994
Title: Comparison of Long-term Results of UGYTEX® Sub-bladder Mesh Placed Via a Transvaginal Transobturator Approach Versus Subvesical Plication Without Reinforcement in the Surgical Treatment of Bladder Prolapse
Brief Title: UGYTEX® Mesh Versus Subvesical Plication in the Surgical Treatment of Bladder Prolapse
Acronym: PRO-CURE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2013/RdeT-01; 2013-A01705-40 (Other: ANSM)
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2016-02

CONDITIONS: Cystocele
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UGYTEX (Experimental): Patients in this arm received the UGYTEX mesh in the pro-cure 1 study (see NCT00153257)
  Interventions: Device: UGYTEX
- No MESH (Active Comparator): Patients in this arm had subvesical plication without reinforcement.
  Interventions: Procedure: No mesh.

INTERVENTIONS:
Device: UGYTEX — Patients in this arm received the UGYTEX mesh in the pro-cure 1 study (see NCT00153257)
  Arms: UGYTEX
Procedure: No mesh. — Patients in this arm had subvesical plication without reinforcement.
  Arms: No MESH

SUMMARY:
The main purpose of this study is to evaluate the long-term (5-8 years) functional prolapse recurrence rate of the 147 patients enrolled, randomized and analyzed in the study PRO-CURE I.

DETAILED DESCRIPTION:
Secondary objectives include comparing the following elements between the two randomized groups at a long-term time point (5-8 years):

A. The anatomic failure rate of cystocele (POP-Q stage > or = 2) B. Late postoperative morbidity C. Residual post-operative pain (visual analog scale (VAS)) D. Patient satisfaction via the PGI-I questionnaire E. Quality of life via the PFDI and PFIQ questionnaires F. Sexual activity via the PISQ-12 questionnaire G. The rate of vaginal erosion H. Displacement and secondary shrinkage of meshs

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient included in, randomized and analysed in the PROCURE study (NCT00153257)

Exclusion Criteria:

* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Patient not included in the PROCURE study

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12-07 (Actual); Study Completion 2015-12-07 (Actual)

PRIMARY OUTCOMES:
Functional failure | 5 years
  The primary efficacy endpoint of this study, is the functional failure at 5 years, defined using the functional response at 12 months in NCT00153257, the concept of surgery for prolapse and the answer to question No. 5 of the PFDI questionnaire submitted between 5 and 8 years postoperatively.

SECONDARY OUTCOMES:
Anatomical failure | 5-8 years
  The anatomical failure is defined by a failure or recurrence at 12 months (data from NCT00153257), or surgery for prolapse or anatomic recurrence (recurrence of cystocele stage 2 or higher) upon examination at 5 to 8 years.
Post-operative complications | 5-8 years
  Major complications include surgery for prolapse repair, re-hospitalization or functional complications. Minor complications include all adverse events that are not major complications. Mesh-specific complications include vaginal pain, vaginal erosions, displacement and retraction of the mesh.
The PGI-I questionnaire | 5-8 years
The PFDI questionnaire | 5-8 years
The PFIQ questionnaire | 5-8 years
The PISQ-12 questionnaire | 5-8 years

CONTACTS AND LOCATIONS:
Overall Officials: Renaud de Tayrac, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (12):
- France (12):
  - Clinique Champeau, Béziers
  - APHP - Hôpital Antoine Beclere, Clamart
  - CHU de Clermont Ferrand - Hôpital Estaing, Clermont-Ferrand
  - APHP - Hôpital Beaujon, Clichy
  - CH d'Issoire - Centre Hospitalier Paul Ardier, Issoire
  - CH de la Rochelle, La Rochelle
  - CH de Chartres - Hôpital Louis Pasteur, Le Coudray
  - APHP - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CH d'Orange - Hôpital Louis Giorgi, Orange
  - Clinique Mutualiste La Sagesse, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen

REFERENCES:
- [Result] Allegre L, Callewaert G, Alonso S, Cornille A, Fernandez H, Eglin G, de Tayrac R. Long-term outcomes of a randomized controlled trial comparing trans-obturator vaginal mesh with native tissue repair in the treatment of anterior vaginal wall prolapse. Int Urogynecol J. 2020 Apr;31(4):745-753. doi: 10.1007/s00192-019-04073-x. Epub 2019 Sep 10. PMID 31506808